CLINICAL TRIAL: NCT05564806
Title: A Multicenter, Open-Label, Phase I Dose Escalation Study To Evaluate The Safety, Tolerability And Pharmacokinetics Of YH004 In Subjects With Advanced Solid Tumors And Relapsed Or Refractory Non-Hodgkin Lymphoma
Brief Title: Study of YH004 (4-1BB Agonist Antibody) in Advanced Solid Tumors And Relapsed Or Refractory Non-Hodgkin Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eucure (Beijing) Biopharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YH004003
Record Dates: First submitted 2022-09-29; First posted 2022-10-04 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2022-10

CONDITIONS: Advanced Solid Tumors; Relapsed Or Refractory Non-Hodgkin Lymphoma

STUDY DESIGN:
Intervention Model Description: Clinical trials with a single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention/treatment (Experimental): All subject will receive YH004 intravenously as single agent every three weeks (Q3W), until intolerable toxicity, disease progression, withdrawal of consent, or Investigator decision, whichever comes first.
  Interventions: Drug: YH004

INTERVENTIONS:
Drug: YH004 — All subject will receive YH004 intravenously as single agent every three weeks (Q3W), until intolerable toxicity, disease progression, withdrawal of consent, or Investigator decision, whichever comes first.

SUMMARY:
This is an multicenter, open-label, dose-escalation study of the study drug YH004 . The study is designed to determine the safety, tolerability, maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of YH004 in subjects with advanced solid tumors and relapsed or refractory Non-Hodgkin lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide signed and dated informed consent prior to any study related procedures and willing and able to comply with all study procedures.
2. Patients with histologically or cytologically confirmed advanced solid tumor or relapsed or refractory Non-Hodgkin Lymphoma (including but not limited to inert and transformed type, patients with inert lymphoma must undergo systematic treatment at the time of screening), which has progressed after treatment with standard therapies or intolerant of standard therapies or have no standard of care.
3. Subject must have at least one measurable lesion by RECIST 1.1 or per Cheson criteria (Lugano 2014).
4. Subjects must be 18 years to 80 years of age at the time of screening.
5. Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Have life expectancy of at least 12 weeks based on investigator's judgement.
7. Sufficient organ and bone marrow functions before screening or administration.
8. Women of reproductive potential must have negative serum beta human chorionic gonadotropin (β -HCG) pregnancy test at the time of screening.
9. Women of reproductive potential who are sexually active must consistently use highly effective contraception/birth control (less than 1% per year) between signing of the informed consent and 90 days after the last administration of the study drug.

Exclusion Criteria:

1. Previous exposure to an anti-CD137 (e.g., utomilumab, urelumab) antibodies.
2. Subjects must not have another active invasive malignancy within 2 years or currently.
3. Subjects have received any anticancer therapy or another investigational agent within the longer of 4 weeks or 5 half-lives before the first dose of the study drug.
4. Continuance of toxicities due to prior anti-tumor therapy that have not recovered to ≤ Grade 1 per CTCAE 5.0.
5. Subjects who have major operations within 4 weeks before the first dose of the study drug, or minor surgery within 2 weeks prior to the first dose.
6. Subjects have received any radiotherapy within the longer of 4 weeks before the first dose of the study drug.
7. Subjects with primary CNS malignancy or symptomatic CNS metastasis.
8. Subjects with a history of ≥ Grade 3 immune-related adverse events resulted from previous immunotherapy or treatment discontinuation due to previous immunotherapy.
9. Subjects must not receive concurrent or prior use of an immunosuppressive agent within 4 weeks of the first dose of study drug.
10. Subjects must not receive any other investigational drug or participated in other clinical studies within 4 weeks before the first dose of study drug.
11. Subjects must not have received a live vaccine or attenuated live vaccine within 4 weeks before the first dose of study drug.
12. Known allergies to the active ingredient or excipients of the test drug, or history of severe allergic reaction (≥ grade 3) to any other monoclonal antibody or intravenous therapeutic protein preparation drug.
13. History of interstitial lung disease or noninfectious pneumonia requiring corticosteroid treatment.
14. More than moderate amount of uncontrollable pleural, abdominal or pericardial effusion requiring repeated drainage or with obvious symptoms.
15. Subjects must not have an active autoimmune disease, a history of autoimmune disease requiring systemic therapy, or a history of autoimmune disease within 2 years of the first dose of study drug.
16. Clinically uncontrolled illness, including but not limited to severe diabetes, uncontrolled hypertension, serious endocrine disorders or other serious diseases requiring systemic treatment such as severe abnormal thyroid function.
17. Subjects must not have a history or persistent active virus or tuberculosis infection. Including but not limited to: human immunodeficiency virus (HIV), syphilis, hepatitis C, hepatitis B or active COVID-19 infection; previous or current active pulmonary tuberculosis and other active infectious diseases.
18. Severe infections requiring intravenous administration within 7 days before the first dose of study drug.
19. Severe cerebro-cardiovascular disease within 6 months of the first dose of study drug, such as cerebrovascular rupture, stroke, myocardial infarction, unstable angina pectoris, congestive heart failure (NYHA grade ≥ II), valvular disease with significant clinical significance, and serious out of control arrhythmia requiring drug treatment (pulmonary hypertension or left ventricular ejection fraction (LVEF) ≤ 50% during screening period).
20. QTc > 480 ms at baseline, corrected for heart rate using Frederica's formula.
21. Subjects must not have a history of allogeneic bone marrow transplantation or organ transplantation.
22. Any known mental illness or disorder, substance abuse history, drug abuse history or alcohol dependence history that would preclude subject from participation.
23. Females who are lactating, except for whom agreed to stop lactating during the trial.
24. Any condition that the investigator believes may not be appropriate for participating the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-10-24 (Estimated); Study Completion 2026-02-07 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | up to 1 year after the last dosing
  The safety profile of YH004 will be assessed by monitoring the adverse events (AE) per NCI CTCAE v5.0.
Maximum tolerated dose (MTD) and/or Recommended phase 2 dose (RP2D) | up to 1 year after the last dosing
  The MTD and/or RP2D will be determined based on the data of safety and tolerability.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang